CLINICAL TRIAL: NCT01201122
Title: Multi Center Ulcerative Colitis Pediatric Pentasa Intervention Trial (MUPPIT). A Randomized, Single-blinded, Controlled, Parallel, Induction Therapy With Once vs. Twice Daily Dosing of Pentasa in Pediatric UC.
Brief Title: Once Versus Twice Daily Mesalamine to Induce Remission in Pediatric Ulcerative Colitis
Acronym: MUPPIT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Arie Levine, Pediatric Gastroenterology and Nutrition Unit, Wolfson Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0052-10-WOMC
Record Dates: First submitted 2010-09-12; First posted 2010-09-14 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Mild to Moderate Ulcerative Colitis
Keywords: Pediatric; Ulcerative colitis; 5-ASA; Mesalamine; Dosing
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Weight based Mesalamine: Once daily (Experimental)
  Interventions: Drug: Mesalamine
- Weight based Mesalamine: Twice daily (Experimental)
  Interventions: Drug: Mesalamine

INTERVENTIONS:
Drug: Mesalamine — Dosing: The current standard of care for pediatric UC is 75mg/kg/day of mesalamine (Pentasa) and should be in multiplications of 500mg (half sachets).
  Patients will be randomized in blocks of six stratified by weight groups: 15- <30 kg, 30-40kg, >40kg.
  For body wt. 15- <20kg Arm: Once daily, 1000 mg (morning) and Placebo (0.5 sachet) (evening). Arm: Twice daily, 500mg (morning) and 500mg (evening).
  For body wt: 20- <30 kg Arm: Once daily, 1500mg (morning) and Placebo (0.5 sachet) (evening). Arm: Twice daily, 1000mg (morning) and 500mg (evening).
  For Body wt. 30- <40 kg Arm: Once daily, 2000mg (morning) and Placebo (1 sachet) (evening). Arm: Twice daily, 1000mg (morning) and 1000mg (evening).
  For body wt. ≥40 kg Arm: Once daily, 3000mg (morning) and Placebo (1.5 sachet) (evening). Arm: Twice daily, 1500mg (morning) and 1500mg (evening).

SUMMARY:
The purpose of this study is to evaluate effectiveness of once daily dosing of Pentasa compared with twice daily in children with mild to moderate active ulcerative colitis.

DETAILED DESCRIPTION:
Several randomized controlled trials (RCTs) have affirmed the efficacy of 5-aminosalicylic acid (5-ASA) and sulfasalazine in the acute treatment of mild to moderate exacerbations, as well as in the maintenance of clinical remission. Initially, common practice was to prescribe 5-ASA in three divided doses. Slow release once daily mesalamine with Multi Matrix System (MMX) technology was shown to be effective in induction and maintenance of remission of adult ulcerative colitis (UC). Since transit time of the colon is much slower than the small-bowel, and since the active ingredient should act locally on the colon, less frequent dosing of the regular formulation may also provide sufficient colonic coverage. Indeed, two recent studies among adults with UC suggest that once daily dosing of mesalamine (Pentasa® and Salofalk®) may be as or more effective than twice daily dosing.

To date, most RCTs have been conducted among adult patients and efficacy in children has been extrapolated from these data. However, childhood inflammatory bowel disease (IBD) may not be similar to adult onset disease. The prevalence of extensive colitis proximal to the splenic flexure is doubled in pediatric-onset UC compared to adults and extensive disease is consistently associated with more severe phenotype. On the other hand, studies in children with IBD often show better response to therapy than in adults. Therefore, American and European regulating agencies encourage pediatric studies be conducted for all approved drug products. It has been found that less than 50% of children with IBD are adherent with treatment, a figure associated with the understanding of the disease which is generally lower than in adults. Therefore, the advantage of once daily dosing of 5-ASA over twice-daily may be greater in children compares with adults.

The investigators hypothesize that once daily dosing of mesalamine is superior in effectiveness to twice daily dosing to induce remission in pediatric mild-moderate UC. We base this hypothesis on data previously found in adults and due to the expected higher adherence rate.

This study will compare two groups receiving an identical dose of the same non experimental medication, with the only difference being in the number of doses of the medication!

ELIGIBILITY:
Inclusion Criteria:

1. Children 6-18 years of age, weight least 15kg.
2. Diagnosis of UC, established by the presence of accepted clinical, radiologic, endoscopic and histologic criteria.
3. Mild to moderate disease activity at the time of enrolment as judged by the Pediatric UC Activity Index (PUCAI) score 10-55 points.
4. In general good health (other than the diagnosis of UC), based on medical history, physical examination, and screening laboratory results.
5. Infectious colitis excluded by stool cultures, ova and parasite examination and Clostridium difficile assay.
6. Ability and acceptance to participate in the study and follow study procedures, as evidenced by a parent/legal guardian signing a written informed consent and the child providing assent.

Exclusion Criteria:

1. Weight <15 kg at enrolment
2. Patients whose disease is confined to the rectum (i.e. proctitis).
3. Fever >38.5 degrees.
4. Patients with Crohn's colitis or with IBD type unclassified (IBD-U) according to Montreal classification.
5. Treatment with oral 5-ASA oral preparation with at least 50mg/kg/day > 3 days within 7 days prior to screening visit. Patients who are treated with 5-ASA <50mg/kg/d may be enrolled as their dose will be increased significantly in this trial. A sensitivity analysis is planned including only 5-ASA naïve children.
6. Exacerbation associated with infectious organism in the stool.
7. Current treatment with steroids (any dose) or the need for steroid therapy as judged by the responsible gastroenterologist.
8. Rectal therapies (suppositories, foams, enemas etc) of all kind are allowed if the dose and frequency has remained stable during the previous 30 days prior to the screening visit. No changes are allowed after randomization and until completion of the study.
9. Treatment with immunomodulatory therapy including, but not limited to: 6 mercaptopurine (6-MP), azathioprine, cyclosporine, tacrolimus, rosiglitazone or methotrexate, is allowed if the dose and frequency has remained stable during the previous 90 days prior to the screening visit. No changes are allowed after randomization and until completion of the study.
10. Treatment with biologic therapy including, but not limited to: infliximab, certolizumab, adalimumab within 90 days prior to screening visit.
11. Pregnancy. All female patients of childbearing potential will undergo urine pregnancy testing at screening, must not be lactating, and willing to use acceptable contraception if sexually active.
12. Known allergy to 5ASA, salicylates, or aminosalicylates.
13. Existence of current renal disease, or a screening blood urea nitrogen (BUN) or creatinine value that is > 1.5 times the upper limit of the age appropriate normal.
14. Existence of current hepatic disease, or liver tests (ALT, AST, T-Bili) that are > 2 times the upper limit of normal, or the existence of Primary Sclerosing Cholangitis (PSC).
15. History of recurrent pancreatitis.
16. Any other laboratory or clinical condition that the investigator considers clinically significant that would impact the outcome of the study or the safety of the patient.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 86 (Actual)
Dates: Start 2010-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Difference in mean PUCAI score between the groups. | At week 6 after initiation of therapy.

SECONDARY OUTCOMES:
Treatment success defined as Complete response OR large partial response. | At 3 and 6 weeks from initiation of therapy.
  Complete response: A a PUCAI score <10 points AND a change of at least 10 points from baseline.
  Small partial response: A a change in PUCAI score of at least 10 points from baseline AND a PUCAI score of ≥10 points.
  Large partial response: A change in PUCAI score of at least 20 points from baseline AND a PUCAI score of ≥10 points.
  Treatment Failure: A lack of improvement of at least 10 points from the baseline PUCAI score despite at least 3 weeks of treatment, or requirement of corticosteroids at any time.

CONTACTS AND LOCATIONS:
Overall Officials: Arie Levine, MD, Study Chair — Pediatric Gastroenterology and Nutrition Unit, The E. Wolfsom MC, Tel-Aviv Universiy, Holon, Israel; Dan Turner, MD, PhD, Study Director — Pediatric Gastroenterology and Nutrition Unit, The Hebrew Universitiy of Jerusalem, Shaare Zedek MC, Jerusalem, Israel; Ron Shaoul, MD, Principal Investigator — Pediatric Gastroenterology Unit, Meyer Children's Hospital, Rambam MC, Haifa, Israel; Batia Weiss, MD, Principal Investigator — Safra Children's Hospital, Sheba MC, Tel-Hashomer, Israel
Locations (1):
- Wolfson Medical Center, Holon, Israel